CLINICAL TRIAL: NCT05534256
Title: Reducing Sedentary Time in Patients With Cardiovascular Disease: A Pilot Randomized Controlled Trial
Brief Title: Reducing Sedentary Time in Patients With Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Chorong Park, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 220416
Record Dates: First submitted 2022-08-24; First posted 2022-09-09 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Sedentary Behavior; Physical Activity
Keywords: Sedentary behavior; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor and statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth.
  Interventions: Behavioral: Sit Less Program
- Control Group (No Intervention): The control group will receive usual medical care and American Heart Association's Healthy Living booklet

INTERVENTIONS:
Behavioral: Sit Less Program — The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth. Outcomes will be measured at baseline and post-intervention
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to develop and test a 12-week sedentary behavior reduction intervention ("Sit Less" program) for patients with cardiovascular disease. The program aims to reduce and break sitting times among this population using an objective activity monitor and mHealth. The investigators will test the program to help cardiovascular disease patients break up sitting time, reduce daily sitting time, and move more. The investigators will also study whether the program leads to improvements in heart disease risk factors, and whether cardiovascular disease patients like the program and can follow it.

DETAILED DESCRIPTION:
The investigators propose to develop and conduct a pilot 2-arm RCT to test a wearable technology-based sedentary behavior reduction intervention in cardiovascular disease patients. Participants will be randomized to either the control group or the sedentary behavior reduction intervention group. The intervention group will target a 120 minute per day reduction in sedentary behavior using an objective activity monitor and mHealth.

Specifically, the study aims to: determine the feasibility and acceptability of the sedentary behavior reduction intervention in cardiovascular patients by evaluating reach, retention, satisfaction, and compliance with the intervention; evaluate the preliminary efficacy of the sedentary behavior reduction intervention on changes in sedentary time; and explore preliminary effects of the sedentary reduction intervention on physical activity, cardiometabolic markers and patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and above
* Have at least one of the following conditions including history of heart attack or peripheral artery disease or a stent placed in heart or leg
* Self-report of sitting ≥ 8 hr/day
* Ability to stand and walk
* Ownership of a smartphone

Exclusion Criteria:

* Currently using an activity tracker
* Currently participating in exercise of cardiac rehabilitation programs
* Non-English speaking
* Patients who are classified as unstable (e.g. heart failure, uncontrolled arrhythmia) or have kidney disease that limits daily water intake, or any other conditions contradictory to standing or walking and
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Level of satisfaction with the intervention assessed by the System Usability Scale and exit-interview | Baseline to 12 weeks
  Level of satisfaction with the intervention will be assessed by using the 10-item of system usability scale. An exit interview will be conducted by the intervention among subsamples of the intervention group (n =20) during the post-intervention visit. The interview will assess the acceptability of and satisfaction with the intervention, barriers and facilitators to sedentary behavior reduction, and any alternate strategies tried by participants during the study.
Level of compliance with the intervention assessed by number of days the Fitbit device was worn | Baseline to 12 weeks
  The compliance with the intervention will be assessed by number of days the Fitbit device was worn per week.
Changes of sedentary behavior assessed by 7 days of activPAL device monitoring | Baseline and 12 weeks
  Sedentary behavior will be assessed by three parameters including total daily sedentary time, prolonged sedentary time (time spent sitting >30mins), and numbers of sit-to-stand transition. These three sedentary behavior parameters will be measured by 7 days of activPAL 3 device monitoring.

SECONDARY OUTCOMES:
Changes of physical activity measured by 7 days of activPAL device monitoring | Baseline and 12 weeks
  Physical activity will be measured by 7 days of activPAL monitoring.
Changes of cardiometabolic biomarkers measured by blood dried spot card | Baseline and 12 weeks
  Cardiometabolic markers including fasting cholesterols, insulin levels, HbA1c, fasting glucose, and hs-CRP will be measured by blood dried spot card. For blood samples, participants will fast overnight (at least 8 hours). The trained RA will conduct a finger prick and 8-9 drops of blood will be obtained on a dried blood spot card.
Changes of confidence in reducing sedentary behavior measured by using 6 items from the Self-Efficacy Questionnaire for Physical Activity and Sedentary Behavior. | Baseline and 12 weeks
  Confidence in reducing sedentary behavior will be measured using 6 items from the Self-Efficacy Questionnaire for Physical Activity and Sedentary Behavior.
Changes of habit strength for sedentary behavior assessed by using the Self-Report Habit Index. | Baseline and 12 weeks
  Habit strength for sedentary behavior will be assessed by 7 items from the Self-Report Sedentary Behavior Habit Index.
Changes of 24-hour glucose levels assessed by continuous glucose monitors | Baseline and 12 weeks
  24-hour glucose levels will be measured by the use of a continuous glucose monitor over a 7-day period. The 24-hour glucose control will be evaluated by mean 24-hour glucose levels and numbers of events and time in hypoglycaemia (glucose < 3.9 mmol/l), euglycaemia (glucose 3.9-7.8 mmol/l), hyperglycaemia (glucose > 7.8 mmol/l) and above target (glucose > 9 mmol/l).

CONTACTS AND LOCATIONS:
Overall Officials: Chorong Park, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
The investigator does not have plans to share data at this time. In the future, reasonable requests for de-identified data from other scientists will be considered. Such data will be shared with approval by the Study PI and other investigators, as appropriate.